CLINICAL TRIAL: NCT02528032
Title: Revisit the Value of Imaging in Best Using CArdiac Resynchronization Therapy
Acronym: RICART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 35RC14-9767
Record Dates: First submitted 2015-08-14; First posted 2015-08-19 (Estimated); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Cardiac Resynchronization Therapy
Keywords: Left ventricular dysfunction; Other cardiac dysrhythmias
MeSH Terms: conditions — Ventricular Dysfunction, Left

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Echocardiographic evaluation (Other): Echocardiographic evaluation of heart function with new processing tools
  Interventions: Other: Echographic evaluation of heart function

INTERVENTIONS:
Other: Echographic evaluation of heart function — Echocardiographic data collection and analysis, not fully exploited at present

SUMMARY:
Many studies have shown the benefits of cardiac resynchronization therapy (CRT) with biventricular pacing in patients with heart failure with left ventricular dysfunction. CRT restores contraction coordination between different regions of the left ventricle, which yields a significant improvement in LV systolic function, symptoms, exercise tolerance and quality of life. In the longer term, treatment with resynchronization induces a reverse remodeling of the left ventricle and a decrease in mortality and morbidity (hospitalization for heart failure). Nevertheless, even if a majority of patients treated with CRT feel the benefit, some (up to 40% depending on the response criteria of CRT) do not experience significant improvement (nonresponders). Echocardiography and imaging have not so far demonstrated their added value to optimize delivery of CRT. Monocentric promising work on limited numbers of patients, however, were carried out. Meanwhile, equipment for delivering CRT evolves and new probes with four poles stimulation of the left ventricle are now used. The objective of this research is to validate new sequences of ultrasound processing estimating the CRT. These tools are based on usual echocardiographic examination of patients

DETAILED DESCRIPTION:
Pilot study for testing tools pre and post-treatment images echocardiography but also MRI with a descriptive purpose and identification of the computed parameters should be secondarily test a large multicenter cohort . Patients in the study will be explored in RICART preimplantation as then in the manner used in current clinical routine. The use of data by cons will focus on the study of new tools ever compared in the same patients.

Data echocardiography (as with other techniques) are those used in clinical routine. Then, the data processing to be carried characterized the asynchrony posteriori, regardless of initial clinical data on a dedicated search software. Each quantitative parameter will be compared with others in order to predict the response to resynchronization. Response prediction of threshold values to the resynchronization can be obtained and compared to each of the tools. The value of relative and an addition to another may be tested.

The predictive value of the change (delta) of each parameter between the pre- and post-implantation to predict response to al resynchronization, will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with sinus rhythm sent to hospital for a cardiac resynchronization according to ESC criteria and implanted with a left ventricular pacing lead quadrupole

Exclusion Criteria:

* Patients with an acoustic window is incompatible with the accurate echographic assessment of heart function
* Patients with spontaneous one year prognosis is not dependent on his heart or another disease to the forefront (eg neoplasia)
* Contra-indications to MRI (pacemaker or implantable defibrillator, intracranial ferromagnetic surgical clips, cochlear implants, intraocular metallic foreign body, Starr-Edwards heart valve prosthesis pre 6000, biomedical device type pump insulin or neurostimulator) or against -indications to iodinated contrast injection (severe renal impairment, allergy).
* Patient not giving free and informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-08; Primary Completion 2018-07 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Measuring the prognostic value of a package of new ultrasonic signal processing tools | pre-implantation
  To evaluate the prognostic value of a package of new tools quantitatively measuring mechanical dyssynchrony prior to implantation of a resynchronization pacemaker in terms of favorable response at 6 months.

SECONDARY OUTCOMES:
Compare pre and post-implantation asynchrony characterisation | pre-implantation, and within three day post implantation
  pre and within three day post implantation mechanical asynchrony by package of new tools will be compared with the same characterization of biventricular pacemaker.
Characterization of the pre-implantation mechanical asynchrony by package of new tools | pre-implantation
  The characterization of the pre-implantation mechanical asynchrony with the package of tested tools will be correlated with the results of:
  * Replacement fibrosis mark (taking gadolinium) and interstitial fibrosis (T1 mapping) [MRI]
  * Evaluation of the coronary venous system by chest CT
Analysis and comparison of cardiac mechanical asynchrony characterization tools with other asynchronism criteria already describe | at 6 month
  cardiac mechanical asynchrony characterization tools will be analyzed and compared, associated with other asynchronism criteria already described defined by the reverse LV remodeling 6 months post-implantation (positive response regressions = ≥15% of tele-systolic volumes VG 6 months) to define the best or the best combination of predictive tools of the response to the CRT)
Prediction score | at 6 month
  definition of a prediction score of the answer to the CRT (echocardiographic and multi-modality)

CONTACTS AND LOCATIONS:
Overall Officials: Erwan Donal, MD/PH/Prof, Principal Investigator — Rennes UH
Locations (1):
- CHU Pontchaillou, Rennes, France

REFERENCES:
- [Result] Galli E, Le Rolle V, Smiseth OA, Duchenne J, Aalen JM, Larsen CK, Sade EA, Hubert A, Anilkumar S, Penicka M, Linde C, Leclercq C, Hernandez A, Voigt JU, Donal E. Importance of Systematic Right Ventricular Assessment in Cardiac Resynchronization Therapy Candidates: A Machine Learning Approach. J Am Soc Echocardiogr. 2021 May;34(5):494-502. doi: 10.1016/j.echo.2020.12.025. Epub 2021 Jan 7. PMID 33422667
- [Result] Aalen JM, Donal E, Larsen CK, Duchenne J, Lederlin M, Cvijic M, Hubert A, Voros G, Leclercq C, Bogaert J, Hopp E, Fjeld JG, Penicka M, Linde C, Aalen OO, Kongsgard E, Galli E, Voigt JU, Smiseth OA. Imaging predictors of response to cardiac resynchronization therapy: left ventricular work asymmetry by echocardiography and septal viability by cardiac magnetic resonance. Eur Heart J. 2020 Oct 14;41(39):3813-3823. doi: 10.1093/eurheartj/ehaa603. PMID 32918449
- [Result] Donal E, Hubert A, Le Rolle V, Leclercq C, Martins R, Mabo P, Galli E, Hernandez A. New Multiparametric Analysis of Cardiac Dyssynchrony: Machine Learning and Prediction of Response to CRT. JACC Cardiovasc Imaging. 2019 Sep;12(9):1887-1888. doi: 10.1016/j.jcmg.2019.03.009. Epub 2019 Apr 17. No abstract available. PMID 31005538
- [Result] Galli E, Hubert A, Le Rolle V, Hernandez A, Smiseth OA, Mabo P, Leclercq C, Donal E. Myocardial constructive work and cardiac mortality in resynchronization therapy candidates. Am Heart J. 2019 Jun;212:53-63. doi: 10.1016/j.ahj.2019.02.008. Epub 2019 Mar 4. PMID 30951976
- [Result] Donal E, Galli E, Cosyns B. Twenty years after starting cardiac resynchronization therapy, do we understand the electromechanical coupling? Eur Heart J Cardiovasc Imaging. 2019 Mar 1;20(3):257-259. doi: 10.1093/ehjci/jey152. No abstract available. PMID 30371762
- [Result] Galli E, Leclercq C, Hubert A, Bernard A, Smiseth OA, Mabo P, Samset E, Hernandez A, Donal E. Role of myocardial constructive work in the identification of responders to CRT. Eur Heart J Cardiovasc Imaging. 2018 Sep 1;19(9):1010-1018. doi: 10.1093/ehjci/jex191. PMID 28954293
- [Result] Galli E, Leclercq C, Fournet M, Hubert A, Bernard A, Smiseth OA, Mabo P, Samset E, Hernandez A, Donal E. Value of Myocardial Work Estimation in the Prediction of Response to Cardiac Resynchronization Therapy. J Am Soc Echocardiogr. 2018 Feb;31(2):220-230. doi: 10.1016/j.echo.2017.10.009. Epub 2017 Dec 13. PMID 29246513